CLINICAL TRIAL: NCT03947463
Title: Pectoral Nerves I, II and Serratus Plane Blocks in Multimodal Analgesia for Mastectomies A Randomized Clinical Trial
Brief Title: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaukat Khanum Memorial Cancer Hospital & Research Centre (Other)
Responsible Party: Principal Investigator, Hammad Najeeb, Fellow in Anesthesia, Shaukat Khanum Memorial Cancer Hospital & Research Centre
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-15-03
Record Dates: First submitted 2019-04-24; First posted 2019-05-13 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Regional Anesthesia
Keywords: Pectoral Nerves I & II block, Serratus Plane Block, General Anesthesia, opioid analgesia, breast cancer and modified radical mastectomy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Registered pain nurse
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PECS block group (Experimental): 20ml of 0.25% bupivacaine was infiltrated between pectoralis major and pectoralis minor muscle and the spread was visualised on the ultrasound screen. similarly, in Serratus plane block, ultrasound probe was placed over the mid-axillary region of the thoracic cage in a sagittal plane. Ribs were identified inferiorly and laterally, until the identification of the 3rd rib in the mid axillary line. 10 ml of 0.25% bupivacaine was infiltrated in between Serratus anterior muscle and Latissimus Dorsi muscle
  Interventions: Procedure: PECS block
- Control group (No Intervention): Patient were given multimodal analgesia without the regional block

INTERVENTIONS:
Procedure: PECS block — After the induction of general anesthesia, PECS block was administered patients via ultrasound guided technique. We used Mindray M7 Portable ultrasound system using linear probe with (5-10 MHz) frequency. After cleaning the infra clavicular and axillary region with 2% chlorhexidine in 70% Alcohol solution, ultrasound probe was placed in the infraclavicular region and pectoral major and minor were identified. After identification of the landmarks, 20 gauge 50mm Visoplex needle was inserted in-plane direction. 20ml of 0.25% bupivacaine (within the safe limit of its dose) was infiltrated between pectoralis major and pectoralis minor muscle and the spread was visualized on the ultrasound screen.
  Arms: PECS block group

SUMMARY:
Acute postoperative pain is a common problem faced by the patient after surgery, most frequently occurring in first 24 hours. Our primary objective was to assess pain score in first 24 hours in PECS block group undergoing mastectomies. Secondary objective was to observe morphine (opioids) and antiemetic consumption in post anesthetic care unit.

DETAILED DESCRIPTION:
Design: Observer Blinded Randomized control trial.

Place and Duration: Department of Anesthesiology, Shaukat Khanum Memorial Cancer Hospital Lahore (SKMCH), from February 2017 to December 2017

Methods: 120 patients more than 18 years, ASA I and II, planned for unilateral elective modified radical mastectomy under general anesthesia were randomly assigned to receive either general anesthesia plus Pectoral Nerve I, II and serratus (PECS) block (n = 60) or general anesthesia alone (n = 60). Pain score at fixed intervals was measured using Numeric Pain Rating Score (NPRS) after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female age 18 or older
* (ASA) I and II
* Scheduled to undergo elective unilateral mastectomy or Modified radical mastectomy (MRM) under general anesthesia.

Exclusion Criteria:

1. Patient's refusal
2. history of allergy to bupivacaine
3. contraindications to regional anaesthesia (coagulopathy and local infection),
4. BMI > 40 kg/m2,
5. patient scheduled for bilateral mastectomies
6. use of chronic pain medications
7. history of illicit drugs or alcohol abuse and history of psychiatric problems.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patient's diagnosed with breast cancer, undergoing mastectomy
Enrollment: 120 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-12-19 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Pain score over 24 hours | First 24 hrs
  Patient's pain intensity was assessed using NPRS (Numeric Pain scoring system). Pain score was assessed at the time of arrival at PACU (0 minute) and then at 30 minutes after surgery and at discharge from PACU. Pain score was then assessed at the surgical floor at 6hours, 12hours and 24hours.

SECONDARY OUTCOMES:
Post operative morphine (opioids) consumption in PACU | first 24 hours
  If the NPRS score was 3 or more, rescue analgesic dose of 1.5 mg of morphine was administered slowly through the IV route and the pain score was reassessed after 15 minutes. If the pain score was still more than 3, additional dose of 1.5 mg morphine was given. This cycle continued till pain resolved.
Antiemetic consumption for treatment of PONV | 120 minutes
  The incidence of PONV was assessed using a 5-point scale (4-0), where 4 was equivalent to vomiting more than once, 3 was equivalent to one episode of vomit, 2 was equivalent to severe nausea, 1 was equivalent to mild nausea and 0 being no nausea. If the PONV score was more than 2, ondansetron 2 mg IV was administered to treat nausea and vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- Shaukat Khanum Memorial Cancer Hospital and Research Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Menhas R, Umer S. Breast Cancer among Pakistani Women. Iran J Public Health. 2015 Apr;44(4):586-7. No abstract available. PMID 26056679
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Andersen KG, Duriaud HM, Jensen HE, Kroman N, Kehlet H. Predictive factors for the development of persistent pain after breast cancer surgery. Pain. 2015 Dec;156(12):2413-2422. doi: 10.1097/j.pain.0000000000000298. PMID 26176893
- [Background] Afonso AM, Newman MI, Seeley N, Hutchins J, Smith KL, Mena G, Selber JC, Saint-Cyr MH, Gadsden JC. Multimodal Analgesia in Breast Surgical Procedures: Technical and Pharmacological Considerations for Liposomal Bupivacaine Use. Plast Reconstr Surg Glob Open. 2017 Sep 15;5(9):e1480. doi: 10.1097/GOX.0000000000001480. eCollection 2017 Sep. PMID 29062649
- [Background] Richebe P, Rivat C, Liu SS. Perioperative or postoperative nerve block for preventive analgesia: should we care about the timing of our regional anesthesia? Anesth Analg. 2013 May;116(5):969-970. doi: 10.1213/ANE.0b013e31828843c9. No abstract available. PMID 23606468
- [Background] Gurkan Y, Aksu C, Kus A, Yorukoglu UH, Kilic CT. Ultrasound guided erector spinae plane block reduces postoperative opioid consumption following breast surgery: A randomized controlled study. J Clin Anesth. 2018 Nov;50:65-68. doi: 10.1016/j.jclinane.2018.06.033. Epub 2018 Jul 2. PMID 29980005
- [Background] Syal K, Chandel A. Comparison of the post-operative analgesic effect of paravertebral block, pectoral nerve block and local infiltration in patients undergoing modified radical mastectomy: A randomised double-blind trial. Indian J Anaesth. 2017 Aug;61(8):643-648. doi: 10.4103/ija.IJA_81_17. PMID 28890559
- [Background] Blanco R. The 'pecs block': a novel technique for providing analgesia after breast surgery. Anaesthesia. 2011 Sep;66(9):847-8. doi: 10.1111/j.1365-2044.2011.06838.x. No abstract available. PMID 21831090
- [Background] Blanco R, Fajardo M, Parras Maldonado T. Ultrasound description of Pecs II (modified Pecs I): a novel approach to breast surgery. Rev Esp Anestesiol Reanim. 2012 Nov;59(9):470-5. doi: 10.1016/j.redar.2012.07.003. Epub 2012 Aug 29. PMID 22939099
- [Background] Porzionato A, Macchi V, Stecco C, Loukas M, Tubbs RS, De Caro R. Surgical anatomy of the pectoral nerves and the pectoral musculature. Clin Anat. 2012 Jul;25(5):559-75. doi: 10.1002/ca.21301. Epub 2011 Nov 28. PMID 22125052
- [Background] Ullah H, Samad K, Khan FA. Continuous interscalene brachial plexus block versus parenteral analgesia for postoperative pain relief after major shoulder surgery. Cochrane Database Syst Rev. 2014 Feb 4;2014(2):CD007080. doi: 10.1002/14651858.CD007080.pub2. PMID 24492959
- [Background] Akram M, Farooqi FM, Irshad M, Faraz Ul Hassan S, Awais SM. Role of addition of Dexamethasone and Ketorolac to lignocaine intravenous regional anesthesia (Bier's Block) to improve tourniquet tolerance and post-operative analgesia in hand and forearm surgery. J Pak Med Assoc. 2015 Nov;65(11 Suppl 3):S128-31. PMID 26878503
- [Background] Shah AA, Rasool A, Alam MA, Naseem Y, Rasool M, Hussain A, Jadoon S, Shah EH, Malik AA, Ahmed N; Salahudin. Efficacy Of Phenylephrine Infusion Verses Colloid Preloading In Resolving Hypotension Due To Spinal Anaesthesia During Caesarean Section. J Ayub Med Coll Abbottabad. 2018 Jul-Sep;30(3):377-380. PMID 30465369
- [Background] Thomas M, Philip FA, Mathew AP, Jagathnath Krishna KM. Intraoperative pectoral nerve block (Pec) for breast cancer surgery: A randomized controlled trial. J Anaesthesiol Clin Pharmacol. 2018 Jul-Sep;34(3):318-323. doi: 10.4103/joacp.JOACP_191_17. PMID 30386013
- [Background] Madabushi R, Tewari S, Gautam SK, Agarwal A, Agarwal A. Serratus anterior plane block: a new analgesic technique for post-thoracotomy pain. Pain Physician. 2015 May-Jun;18(3):E421-4. PMID 26000690
- [Background] Tighe SQ, Karmakar MK. Serratus plane block: do we need to learn another technique for thoracic wall blockade? Anaesthesia. 2013 Nov;68(11):1103-6. doi: 10.1111/anae.12423. Epub 2013 Sep 14. No abstract available. PMID 24032664
- [Background] Naja MZ, Ziade MF, Lonnqvist PA. Nerve-stimulator guided paravertebral blockade vs. general anaesthesia for breast surgery: a prospective randomized trial. Eur J Anaesthesiol. 2003 Nov;20(11):897-903. doi: 10.1017/s0265021503001443. PMID 14649342
- [Background] Terheggen MA, Wille F, Borel Rinkes IH, Ionescu TI, Knape JT. Paravertebral blockade for minor breast surgery. Anesth Analg. 2002 Feb;94(2):355-9, table of contents. doi: 10.1097/00000539-200202000-00023. PMID 11812698
- [Background] Coveney E, Weltz CR, Greengrass R, Iglehart JD, Leight GS, Steele SM, Lyerly HK. Use of paravertebral block anesthesia in the surgical management of breast cancer: experience in 156 cases. Ann Surg. 1998 Apr;227(4):496-501. doi: 10.1097/00000658-199804000-00008. PMID 9563536
- [Background] Lonnqvist PA, MacKenzie J, Soni AK, Conacher ID. Paravertebral blockade. Failure rate and complications. Anaesthesia. 1995 Sep;50(9):813-5. doi: 10.1111/j.1365-2044.1995.tb06148.x. PMID 7573876